CLINICAL TRIAL: NCT05983302
Title: Repairing Gel (Supraz) and Platelet-rich Plasma-Fibrin Glue (PRP-FG) in Eliminating Odor and Healing the Malodorous Chronic Wounds Versus Standard of Care
Brief Title: Elimination of Odor and Treatment of Malodorous Recalcitrant Wounds by Using Supraz and PRP-FG Versus Standard of Care
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Daryoush Hamidi Alamdari, PhD, Associate professor, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: IR.MUMS.REC.1402.089
Record Dates: First submitted 2023-06-30; First posted 2023-08-09 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Wounds and Injuries
Keywords: Platelet-Rich Plasma-Fibrin Glue; Repairing Gel; Chronic Wounds; Malodorous; Recalcitrant
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Platelet-Rich Plasma-Fibrin Glue (Experimental): The first intervention group (group A) includes 10 patients with chronic wounds who, despite classic wound irrigation treatment, will be undergoing platelet-rich plasma-fibrin glue intervention for 8 weeks.
  Interventions: Drug: Platelet-Rich Plasma-Fibrin Glue
- Repairing Gel (Experimental): The second intervention group (group B) includes 10 patients with chronic wounds who, despite classic wound irrigation treatment, will be undergoing repairing gel intervention for 8 weeks. The components of repairing gel are vitamin A - vitamin C - vitamin B3 - glycine amino acid. - ethanol - collagen - citric acid - glycerin - malic acid - urea - carboxymethyl cellulose - Sodium alginate - Benzoic acid - Allantoin - Bromelain - Methylene blue - Violet dimethyl sulfoxide . The formulation is patented. (PCT, IR108458)
  Interventions: Drug: Repairing Gel
- Platelet-Rich Plasma-Fibrin Glue and Repairing Gel (Experimental): The third intervention group (group C) includes 10 patients with chronic wounds who, despite classic wound irrigation treatment, will be undergoing the repairing gel with approved wound healing components and platelet-fibrin glue for 8 weeks.
  Interventions: Drug: Repairing Gel and Platelet-Rich Plasma-Fibrin Glue
- Classical wound irrigation (control) (Experimental): For 10 patients with chronic wounds, only classical wound irrigation by normal saline (0.9%) will be continued for 8 weeks.
  Interventions: Other: Classical wound irrigation (control)

INTERVENTIONS:
Drug: Platelet-Rich Plasma-Fibrin Glue — The first intervention group includes 10 patients with chronic wounds who, despite common treatment, will be undergone PRP-FG intervention for 8 weeks.
  Other Names: PRP-FG
  Arms: Platelet-Rich Plasma-Fibrin Glue
Drug: Repairing Gel — The second intervention group includes 10 patients with chronic wounds who, despite common treatment, will be undergone the repairing gel with approved wound healing components in the form of gel for 8 weeks.
  Other Names: Supraz Gel
  Arms: Repairing Gel
Drug: Repairing Gel and Platelet-Rich Plasma-Fibrin Glue — The third intervention group includes 10 patients with chronic wounds who, despite common treatment, will be undergone the repairing gel with approved wound healing components in the form of gel and PRP-FG for 8 weeks.
  Other Names: Supraz Gel and PRP-FG
  Arms: Platelet-Rich Plasma-Fibrin Glue and Repairing Gel
Other: Classical wound irrigation (control) — For 10 patients with chronic wounds, only the classical wound irrigation by normal saline will be continued for 8 weeks.
  Other Names: Control
  Arms: Classical wound irrigation (control)

SUMMARY:
The aim of this study is to eliminate the malodorous of chronic wound and increase the chance of the healing of recalcitrant wounds by using the repairing gel (supraz gel) which has the approved components in wound healing and platelet-rich plasma-fibrin glue.

DETAILED DESCRIPTION:
The current study assesses the effects of platelet-rich plasma-fibrin glue (PRP-FG) along with the use of the repairing gel which has the approved components on wound healing in patients with chronic wounds and to eliminate the malodorous of chronic wound. This randomized controlled trial is performed on patients with chronic wounds. Patients will be treated with repairing gel (supraz gel) plus PRP-FG dressing (intervention group) or only Supraz gel (intervention group) or only PRP-FG dressing (intervention group) every 48 hours for 8 weeks versus standard of care of treatment (control group: irrigation of wound by normal saline 0.9%).

ELIGIBILITY:
Inclusion Criteria:

* Having a single wound on the body that has been at least 3 months old and has not been repaired by wound irrigation with normal saline and changing the dressing
* Having a body mass index of 18-35
* Sign the informed consent by the patient

Exclusion Criteria:

* Having concurrent diseases that may cause problems in wound healing, such as cancers, vasculitis, kidney and liver failure, and heart failure
* Taking certain drugs that may interfere with wound healing, such as corticosteroids, immunosuppressive agents, and cytotoxic agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
Wound Odor Change | At the beginning of the study (0 day) and at the end of the eighth week of the intervention (8 weeks)
  Change from Baseline Wound Odor intensity at 2 months will be assessed by the nurse using a Visual Analog Scale (VAS) from 0 to 100 (perceived odor).
Wound Size Change | At the beginning of the study (0 day) and at the end of the eighth week of the intervention (8 weeks)
  Change from Baseline Wound Size (length and width) at 2 months will be assessed in digital images taken of the wound.
Visual Analog Scale changes for pain assessment | Every 48 hours for 8 weeks
  Pain will be evaluated by the visual analog scale system (VAS) which assesses changes in pain via a continuous measurement instrument. The score is determined by measuring the distance (mm) between the no-pain anchor to the point that the patient marks, providing a range of scores from 0 - 10. A higher score indicates greater pain intensity.
Duration of recovery | 8 weeks
  The duration of recovery, which is the number of days it will be taken for the wound to heal.
Change in the systemic inflammatory marker C-reactive protein (CRP) | At the beginning of the study (0 day) and at the end of the eighth week of the intervention (8 weeks)
  C-reactive protein (CRP)
Change in systemic inflammatory marker erythrocyte sedimentation rate (ESR) | At the beginning of the study (0 day) and at the end of the eighth week of the intervention (8 weeks)
  erythrocyte sedimentation rate (ESR)
Change in systemic inflammatory marker Interleukin 6 (IL-6) | At the beginning of the study (0 day) and at the end of the eighth week of the intervention (8 weeks)
  Interleukin 6 (IL-6)
Number of participants with infection | At the beginning of the study (0 day) and at the end of the eighth week of the intervention (8 weeks)
  A swab culture: Identify a small area (1 cm) of clean viable tissue and rotate the swab on it for 5 seconds while applying enough pressure to produce exudate and culture it to detect bacteria.
Results of the SF36 questionnaire at inclusion | Day 0
  The SF-36 questionnaire is a quality-of-life questionnaire that includes 36 questions divided into 8 different categories (physical functioning, limitations due to physical condition, physical pain, perceived health, vitality, social functioning or well-being, limitations due to mental condition, mental health). These 8 dimensions are used to calculate two scores on the quality of life of individuals: the physical composite score and the mental composite score. The higher the score, the greater the capacity. It is self-administered and takes less than 10 minutes. Higher scores indicate better quality of life. The French version has been validated and has satisfactory psychometric properties. Score from 0 to 100.
Results of the SF36 questionnaire at Month 2 | Month 2
  The SF-36 questionnaire is a quality-of-life questionnaire that includes 36 questions divided into 8 different categories (physical functioning, limitations due to physical condition, physical pain, perceived health, vitality, social functioning or well-being, limitations due to mental condition, mental health). These 8 dimensions are used to calculate two scores on the quality of life of individuals: the physical composite score and the mental composite score. The higher the score, the greater the capacity. It is self-administered and takes less than 10 minutes. Higher scores indicate better quality of life. The French version has been validated and has satisfactory psychometric properties. Score from 0 to 100.

SECONDARY OUTCOMES:
Percentage rate of re-epithelialization | Participants will be followed for the duration of 8 weeks
  Pictures taken of the wound site every other day will be analyzed using imaging software for the size of the wound. The percentage rate will be calculated from this.

CONTACTS AND LOCATIONS:
Overall Officials: Daryoush Hamidi Alamdari, Ph.D, Principal Investigator — Surgical Oncology Research Center, Mashhad University of Medical Sciences, Mashhad, Iran.; George Koliakos, MD, PhD, Principal Investigator — Medical School, Aristotle University of Thessaloniki, Thessaloniki, Greece.
Locations (2):
- Medical School, Aristotle University of Thessaloniki, Thessaloniki, Greece
- Mashhad University of Medical Sciences, Mashhad, Razavi Khorasan Province, Iran

IPD SHARING:
Plan to Share IPD: Yes
All data related to the project after the unidentifiable people will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Access to data is allowed 6 months after the publication of results.
Access Criteria: The investigator's data will be available to university staff and academic institutions.